CLINICAL TRIAL: NCT05218876
Title: Effects of Moderate and High-Intensity Exercise During (Neo-)Adjuvant Chemotherapy on Muscle Cellular Outcomes in Women With Breast Cancer: a Randomized Controlled Trial
Brief Title: Effects of Moderate and High-intensity Exercise During Chemotherapy on Muscle Cells in Women With Breast Cancer
Acronym: PhysCan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Norwegian Cancer Society (Other); University of Agder (Other); Haukeland University Hospital (Other); Uppsala University (Other); Active against Cancer - Norway (Unknown)
Responsible Party: Principal Investigator, Truls Raastad, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PhysCan muskel
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Female
Keywords: Muscle fiber cross-sectional area; Muscle biopsies; Training; Oncology; Strength training; Endurance training
MeSH Terms: conditions — Neoplasms | interventions — Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person performing all analyses on muscle tissue (primary outcome) is masked for intervention applied to the individuals and timepoint. The person doing the physical test is not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low- to moderate intensity strength and endurance training (Experimental): Participants will perform a combination of strength and endurance training with low-to moderate-intensity during (neo-) adjuvant treatment with chemotherapy, approximately 6 months. All strength training will be supervised while the endurance training is home-based and followed up by a coach.
  Interventions: Other: Low- to moderate intensity strength and endurance training
- High intensity strength and endurance training (Experimental): Participants will perform a combination of strength and endurance training with high intensity during (neo-) adjuvant treatment with chemotherapy, approximately 6 months. All strength training will be supervised while the endurance training is home-based and followed up by a coach.
  Interventions: Other: High intensity strength and endurance training

INTERVENTIONS:
Other: Low- to moderate intensity strength and endurance training — Combination of strength and endurance training with low- to moderate intensity during chemotherapy
  Arms: Low- to moderate intensity strength and endurance training
Other: High intensity strength and endurance training — Combination of strength and endurance training with high intensity during chemotherapy
  Arms: High intensity strength and endurance training

SUMMARY:
(Neo-)adjuvant chemotherapy for breast cancer has deleterious effects on muscle tissue resulting in reduced skeletal muscle mass, muscle function, and cardiorespiratory fitness. Various exercise regimens during cancer treatment have been shown to counteract some of these side effects. However, no study has compared the effect of high intensity training vs. low-to moderate intensity training on muscle tissue cellular outcomes and function in breast cancer patients during chemotherapy. The present study aims to compare the effects of high vs. low-to moderate intensity training on its ability to counteract deleterious effects of chemotherapy on skeletal muscle in women diagnosed with breast cancer. Eighty newly diagnosed women with breast cancer planned to start (neo-)adjuvant chemotherapy will be randomized to either a group performing a combination of strength and endurance training with high intensity or a group performing training with low to moderate intensity. Muscle biopsies from m. vastus lateralis for assessment of muscular cellular outcomes will be collected and muscle function and cardiorespiratory fitness will be measured before the first cycle of chemotherapy (or, when not possible, one week after) (T0), halfway through chemotherapy (T1), and after completion of chemotherapy (T2). It is estimated that approximately 50% will be willing to take muscle biopsies. The study will give important information about the effects of different training intensities for breast cancer patients during treatment and will contribute with knowledge about how to refine exercise programs that are effective and compatible with multidisciplinary management of breast cancer.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects high and low-to-moderate exercise intensity on muscle cellular outcomes, muscle function, and cardiorespiratory fitness in breast cancer patients undergoing (neo-)adjuvant chemotherapy. We further aim to investigate if treatment including taxane treatment have larger negative effect on muscle than taxane-free treatment.

Our hypotheses are:

* Both high-intensity and low to moderate intensity strength and endurance training during (neo-)adjuvant chemotherapy will reduce negative treatment effects on muscle fiber size, mitochondrial function, cellular stress, and thus reduce the negative effect on cardiorespiratory fitness and muscle function. High-intensity training will be superior to low to moderate-intensity training in counteracting the negative treatments effects.
* Both high-intensity and low to moderate intensity strength and endurance training during (neo-)adjuvant chemotherapy will increase muscle and blood levels of potential anti-tumor myokines.
* Treatment including taxane administration will have larger negative effect on muscle fiber size, mitochondrial function, cellular stress, and thus cardiorespiratory fitness and muscle function than taxane free treatment regardless of training intensity.

This study is a two-group randomized controlled trial. The participants will be randomly allocated into two training groups; one group performing the combination of strength and endurance training with high intensity and the other group performing the training with low to moderate intensity during (neo-) adjuvant treatment for breast cancer. Power calculations indicate that 20 participants are sufficient in each group for our primary outcome muscle fiber cross-sectional area. As we estimate that approximately 50% of the participants will be willing to take muscle biopsies a total of 80 participants will be recruited leading to a total of 40 participants with muscle biopsies.

Before the training period (T0) muscle biopsies, questionnaires and blood samples will be taken before the first chemotherapy cure. The first 2-4 weeks after cure 1 will be used as a familiarization period for tests and exercises, and to complete the remaining T0 tests. Testing will include measurements of physical capacity, body composition, and physical activity levels. All measurements are repeated halfway into the treatment (T1) and after the completion of treatment (T2). Training will start between cures 2 and 3 and will last throughout the treatment period, approximately 6 months.

The strength training consists of two supervised sessions per week and includes the following exercises: seated leg-press, chest-press, seated leg-curl, seated-row, leg-extension, and standing overhead-press using dumbbells. The low-to-moderate intensity group will perform 12 repetitions for 3 sets at 50% of 6RM load in the first weekly session and 20 repetitions for 3 sets at 50% of 10RM load in the second weekly session. The high intensity group will perform 6 repetitions for 3 sets at 6RM load in the first weekly session and 10 repetitions for 3 sets at 10RM load in the second weekly session.

The endurance exercise is home-based and followed up by a coach. The low-to-moderate intensity group do continuous-based exercise (running, cycling, walking uphill or any other endurance-based activity) in bouts of at least 10 min at an exercise intensity of 40-50% of the heart rate reserve. The exercise frequency is recommended to be 2-4 times a week with the main aim to reach 150 min of moderate intensity endurance exercise per week. The high intensity group conduct high-intensity interval exercise. The sessions will consist of two-minute exercise intervals (running, cycling, walking uphill or any other endurance-based activity) at an exercise intensity of 80-90% of the heart rate reserve (at the end of the 3rd session) with two minutes of rest between intervals. During the first week after familiarization, each session will consist of 6 intervals. Thereafter, one bout will be added every fourth week until 10 bouts per session are reached as the maximum, corresponding to 75 min of high intensity per week.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stage I-III breast cancer
* 18 years old
* can understand and communicate in the Norwegian language
* scheduled to undergo (neo-)adjuvant chemotherapy with a combination of taxanes and anthracyclines or only one of the treatments

Exclusion Criteria:

* unable to perform basic activities of daily living
* cognitive disorders or severe emotional instability
* other disabling comorbidities that might hamper physical training (e.g. severe heart failure, chronic obstructive pulmonary disease, orthopedic conditions, and neurological disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Muscle fiber cross-sectional area | From baseline (T0) to the 6 months time point (end of treatment and training, T2)
  Change from baseline (T0) to end of intervention (end of training and treatment), approximately 6 months (T2) in muscle fiber cross-sectional area. This will be assessed by immunohistochemical staining of muscle fiber cross-sections for type 1 and type 2 muscle fibers and dystrophin (cell border).

SECONDARY OUTCOMES:
Muscle fiber cross-sectional area | From baseline (T0) to the 3 months time point (halfway into the treatment and training,T1)
  Change from baseline (T0) to halfway into the intervention (halfway into training and treatment), approximately 3 months (T1) in muscle fiber cross-sectional area. This will be assessed by immunohistochemical staining of muscle fiber cross-sections for type 1 and type 2 muscle fibers and dystrophin (cell border).
Satellite cell content in muscle fiber cross-sections | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in satellite cell content in muscle fiber cross-sections. This will be assessed through immunohistochemical staining of satellite cells in muscle fiber cross-sections for type 1 and type 2 muscle fibers separately.
Myonuclei content in muscle fiber cross-sections | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in myonuclei content in muscle fiber cross-sections. This will be assessed through immunohistochemical staining of myonuclei in muscle fiber cross-sections for type 1 and type 2 muscle fibers separately.
Protein levels of regulators of muscle fiber size (proteins involved in muscle protein synthesis and protein degradation (e.i. mTOR, MuRF, S6K1, p70S6k) | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in protein levels of regulators of muscle fiber size (proteins involved in muscle protein synthesis and protein degradation [e.i. mTOR, MuRF, S6K1, p70S6k]). This will be assessed in muscle homogenate using Western blot analysis.
Protein levels of regulators of muscle fiber cellular stress (Heat Shock proteins: Hsp 27, αB-crystalline, Hsp 60 and Hsp 70) | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in protein levels of regulators of muscle fiber cellular stress (Heat Shock proteins: Hsp 27, αB-crystalline, Hsp 60 and Hsp 70). This will be assessed in muscle homogenate using Western blot analysis.
Protein levels of regulators of mitochondrial function (Citric syntase, Cox 4 and HADH) | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in protein levels of regulators of mitochondrial function (Citric syntase, Cox 4 and HADH). This will be assessed in muscle homogenate using Western blot analysis.
Myokines with potential anti-tumor effects | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in myokines with potential anti-tumor effects. This will be assessed in muscle homogenate using Western blot analysis.
Maximal muscle strength | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in maximal upper- and lower extremity muscle strength. This will be assessed as one repetition maximum in seated chest-press, seated single-leg press and knee extension.
Cardiorespiratory fitness | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in cardiorespiratory fitness. This will be assessed as maximal oxygen uptake during maximal walking/running until exhaustion on a treadmill.
Muscular endurance | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in muscular endurance. This will be assessed as the number of repetitions on 30% of one-repetition maximum in knee extension.
Fat free mass | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in fat free mass. This will be asses by dual dual energy X ray absorptiometry.
Fat mass | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in fat mass. This will be asses by dual dual energy X ray absorptiometry.

OTHER OUTCOMES:
Blood lipids | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in blood lipids. This will be assessed in blood serum and plasma using ELISA methods.
C-reactive protein | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in C-reactive protein. This will be assessed in blood serum and plasma using ELISA methods.
Creatine kinase | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in creatine kinase. This will be assessed in blood serum and plasma using ELISA methods.
Blood glucose | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in blood glucose. This will be assessed in blood serum and plasma using ELISA methods.
Cortisol | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in cortisol. This will be assessed in blood serum and plasma using ELISA methods.
Hemoglobin | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in hemoglobin. This will be assessed in whole blood using standard clinical measures.
Physical activity, defined as minutes spent in moderate-to-vigorous intensity activity | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in physical activity. This will be assessed by the SenseWear Armband activity monitoring device. A SenseWear Armband is worn for 7 consecutive days each time point.
Fatigue | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in fatigue. This will be assessed using the Multi Dimensional Fatigue Inventory (MFI).
Quality of life assessed using EORTC-QLQ30 | From baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2)
  Change from baseline (T0) to the 3 months time point (T1) and from baseline to the 6 months time point (T2) in quality of life. This will be assessed using The European Organization for Research and Treatment of Cancer (EORTC)EORTC-QLQ30.

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, Professor, Principal Investigator — Department of Physical Performance, Norwegian School of Sports Science
Locations (1):
- Haukeland University Hospital, Bergen, Vestlandet, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vikmoen O, Wiestad TH, Thormodsen I, Nordin K, Berntsen S, Demmelmaier I, Strandberg E, Raastad T. Effects of High and Low-To-Moderate Intensity Exercise During (Neo-) Adjuvant Chemotherapy on Muscle Cells, Cardiorespiratory Fitness, and Muscle Function in Women With Breast Cancer: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Nov 11;11(11):e40811. doi: 10.2196/40811. PMID 36367769